CLINICAL TRIAL: NCT02324933
Title: Post-Operative Pain Control in Opioid Tolerant Patients: Fentanyl Challenge Protocol Versus Standard of Care
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: insufficient population, unable to recruit
Sponsor: Bassett Healthcare (Other)
Responsible Party: Principal Investigator, Jose Raul Monzon, M.D., Attending physician - general surgery, Bassett Healthcare
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1064
Record Dates: First submitted 2014-12-19; First posted 2014-12-24 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2015-10

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Fentanyl; Midazolam

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fentanyl Challenge Dosing (Experimental): In the operating room a fentanyl infusion will be started at 2 mcg/kg/min. The time from start of the infusion to respiratory depression(rate < 5 breaths/minute) will be used to calculate the effect-site concentration (Ce).Using the pharmacodynamic model calculated by the Stanpump PCA software, the infusion will continue intraoperatively to achieve a fentanyl Ce of 30%. In the Post Anesthesia Care Unit (PACU), the rate would be changed with the following parameters:
  1. 50% of the hourly dose is given as a basal infusion
  2. The remainder of the hourly dose is ordered as a demand dose q 15 minutes. Post-operatively, the basal rate is adjusted according to the average demand dose use. In patients using < 1 demand dose per hour, the basal rate is decreased by 20%. In patients using > 3 demand doses per hour, the basal rate is increased by 20%. Patients whose pain cannot be managed by this protocol will be removed from the study and pain management will revert to the primary service.
  Interventions: Drug: Fentanyl
- Standard of Care (Control) (Active Comparator): Patients in the best practice arm would receive pre-operative sedation in the operating room comparable to the dose normally given in the Ambulatory Surgery Unit as a "simulated fentanyl challenge". Best practice (control) patients will be followed by the Pain & Palliative Care team in order to make adjustments in pain management as required by the patients.
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Fentanyl — Fentanyl Patient Controlled Analgesia for post-operative pain management
  Other Names: Versed

SUMMARY:
This study will evaluate the value of dosing pain medications based upon a patient's pre-operative tolerance to pain medications. Study participants will be assigned to one of two groups, a treatment group and a control group. The treatment group will be given pain medications after surgery based upon their measured response to pain medications prior to surgery. The control group will be given pain medications based upon the normal dosing routine as is currently practiced. Both groups will be closely monitored for side effects and have their pain scores recorded for the first 48 hours following surgery.

DETAILED DESCRIPTION:
This study will focus on patients who are opioid-tolerant pre-operatively, a patient population which typically has both higher pain scores and more complications related to analgesics than opioid naïve patients. Currently, there is no standardized system for determining an adequate pain control regimen for a patient post-operatively. At this institution, pain medications are dosed per physician preference. The most widely-discussed method for calculating tolerance to opioids relies on converting a patient's daily opioid consumption to a morphine equivalent dose and basing a pain regimen upon that number. This method does not account for variability of response to different medications or dosing forms however. It would be advantageous to have a method of dosing opioid pain medications in this population that is both safe and effective.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18
2. Anticipated need for PCA dosing post-operatively
3. Will undergo major general, plastic, vascular, thoracic or spine surgery
4. Have taken opioid medications orally or transdermally daily for the past 30 days

Exclusion Criteria:

1. Patients assessed to have a difficult airway
2. Known sensitivity or allergy to fentanyl

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-08; Primary Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Pain Score | 48 hours post-operatively
  Patients will rate their pain on a scale of 1-10 (1 being best, 10 being worst)

SECONDARY OUTCOMES:
Pain Score | 24 hours post-operatively
  Patients will rate their pain on a scale of 1-10 (1 being best, 10 being worst)
Events requiring intervention for respiratory depression | 48 hours post-operatively
  All adverse events will be documented including administration of naloxone, prompting to take more frequent breaths by staff and respiratory rate less than 8 per minute
Number of dose adjustments required | 48 hours post-operatively
  Study will record the number of dose adjustments required to maintain adequate pain control

CONTACTS AND LOCATIONS:
Overall Officials: jose Monzon, MD, Principal Investigator — Bassett Healthcare
Locations (1):
- Bassett Healthcare Network, Cooperstown, New York, United States

REFERENCES:
- [Background] Davis JJ, Swenson JD, Hall RH, Dillon JD, Johnson KB, Egan TD, Pace NL, Niu SY. Preoperative "fentanyl challenge" as a tool to estimate postoperative opioid dosing in chronic opioid-consuming patients. Anesth Analg. 2005 Aug;101(2):389-395. doi: 10.1213/01.ANE.0000156563.25878.19. PMID 16037150